CLINICAL TRIAL: NCT03415633
Title: Validity and Cost-effectiveness Analysis of a Home Respiratory Polygraphy for the Diagnosis of Obstructive Sleep Apnea
Brief Title: Validity of a Home Respiratory Polygraphy for the Diagnosis of Obstructive Sleep Apnea
Acronym: APNiA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Araba (Other)
Collaborators: BTI Biotechnology Institute S.L (Unknown); Instituto de Investigación Sanitaria BIO-ARABA (Unknown)
Responsible Party: Principal Investigator, Joaquin Duran-Cantolla, MD, Principal Investigator. MD, PhD, Hospital Universitario Araba
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015-026
Record Dates: First submitted 2016-09-30; First posted 2018-01-30 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: Home Respiratory Polygraphy; Standard Polysomnography; Validity; Cost-effectiveness
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Reproducibility of Results

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Diagnostic Randomizing (Active Comparator): Randomizing to start with home respiratory polygraphy (APNIA) or Standard Polysomnography (PSG)
  Interventions: Other: Home Respiratory Polygraphy (APNIA); Other: Standard Polysomnography (PSG)
- Therapeutic Randomizing (Active Comparator): Randomizing for therapeutic decision taken with home respiratory polygraphy (APNIA) or Standard Polysomnography (PSG)
  Interventions: Other: Home Respiratory Polygraphy (APNIA); Other: Standard Polysomnography (PSG)

INTERVENTIONS:
Other: Home Respiratory Polygraphy (APNIA) — Randomizing to start with home respiratory polygraphy (APNIA)
  Other Names: Validity
  Arms: Diagnostic Randomizing
Other: Standard Polysomnography (PSG) — Randomizing to start with Standard Polysomnography (PSG)
  Other Names: Validity
  Arms: Diagnostic Randomizing
Other: Home Respiratory Polygraphy (APNIA) — Randomizing for therapeutic decision taken with home respiratory polygraphy (APNIA)
  Other Names: Effectiveness
  Arms: Therapeutic Randomizing
Other: Standard Polysomnography (PSG) — Randomizing for therapeutic decision taken with Standard Polysomnography (PSG)
  Other Names: Effectiveness
  Arms: Therapeutic Randomizing

SUMMARY:
To assess the diagnostic validity and cost-effectiveness of a APNiA device, a home respiratory polygraphy (HRP).

DETAILED DESCRIPTION:
To assess the diagnostic validity and cost-effectiveness of a APNiA device, a home respiratory polygraphy (HRP), performed at home compared with the standard polysomnography (PSG) in adults with clinically suspected Obstructive Sleep Apnea (OSA).

METHODOLOGY: DESIGN: Randomized, prospective, multicenter, and crossover trial. The study will include 240 adults, both sexes, with clinical suspicion of obstructive sleep apnea (OSA). MEASUREMENTS: To all patients with clinical suspected OSA and referred to the sleep units, the following questionnaires and measurements will be performed: a) clinical history; b) Anthropometric variables: weight, height, body mass index, neck circumference and percentile; c)Epworth sleepiness scale; OSA questionnaire, quality of life and clinical questionnaires and comorbidity; d) PSG in the sleep laboratory; e) HRP at home; f) Cost-effectiveness variables.

ANALYSIS: Data from HRP and from full PSG will be compared as follows: 1) Agreement of results according to the different apnea-hypopnea index by using the Receiver Operating Characteristic (ROC) curve; 2) The concordance of the diagnosis and treatment decisions when using clinical findings and data from PSG or HRP at home; 3) All data will be analyzed independently; 4) A cost-effectiveness analysis of the different diagnostic and therapeutic procedures will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years to 75 years old, with clinical suspicion of OSA
* Written informed consent signed

Exclusion Criteria:

* Psycho-Physical inability to perform the study at home
* Presence of insomnia or depressive syndrome
* Patient with malformation syndromes, Down syndrome and neuromuscular diseases
* Cardiovascular, cerebrovascular or respiratory disease exacerbated.
* Previous Positive continuous pressure (CPAP ) treatment or surgery for OSA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2015-09; Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | baseline
  To assess the diagnostic validity of a home respiratory polygraphy (HRP) compared with the standard polysomnography (PSG) in adults with clinically suspected Obstructive Sleep Apnea (OSA), based on the results of the Apnea-hypopnea Index (AHI).

SECONDARY OUTCOMES:
Therapeutic decision | 6 month
  The concordance of the diagnosis and treatment decision when using clinical findings and data from standard polysomnography (PSG) or home respiratory polygraphy (HRP).
Epworth Sleepiness Scale | baseline and at 6 month
  The Epworth Sleepiness Scale (the sum of 8 items score,0-3) can range from 0 to 24. Scores of 11-24 represent increasing levels of excessive daytime sleepiness.
STOP-BANG Sleep apnea questionnaire | baseline and at 6 month
  Sleep Apnea Questionnaire. High STOP-Bang score indicates a high probability of obstructive sleep apnea.
Berlin questionnaire | baseline and at 6 month
  The questionnaire consists of 3 categories related to the risk of having sleep apnea. Patients can be classified into High Risk or Low Risk based on their responses to the individual items and their overall scores in the symptom categories.
  High Risk:
  if there are 2 or more categories where the score is positive.
  Low Risk:
  if there is only 1 or no categories where the score is positive.
Cost-effectiveness analysis | 6 month
  Cost-efficacy evaluation
Blood pressure | baseline and at 6 month
  Blood pressure measurements: systolic blood pressure and diastolic blood pressure
Anthropometric variables (Body mass index) | baseline and at 6 month
  Body mass index
Quality of life (EuroQOL test) | baseline and at 6 month
  Evaluate by EuroQOL test, is a standardised measure of health status. Description of the state of health in five dimensions (mobility, self-car, usual activities, pain/discomfort and anxiety/depression), each o wich is defined with three levels of severity, as measured by a Likert scale type (no problems, some problems and many problems or inability to activity).

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Duran-Cantolla, Study Director — Hospital Universitario Araba; Eduardo Anitua-Aldecoa, Principal Investigator — BTI Technology Institute SL
Locations (1):
- Hospital Universitario Araba, Vitoria-Gasteiz, Araba, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Durán-Cantolla J, Puertas FJ, Pin G y el Grupo Español de Sueño (GES).Documento de consenso nacional sobre el SAHS. Arch Bronconumol 2005;41(nº4):1-110.
- [Background] Lloberes P, Duran-Cantolla J, Martinez-Garcia MA, Marin JM, Ferrer A, Corral J, Masa JF, Parra O, Alonso-Alvarez ML, Teran-Santos J. Diagnosis and treatment of sleep apnea-hypopnea syndrome. Spanish Society of Pulmonology and Thoracic Surgery. Arch Bronconeumol. 2011 Mar;47(3):143-56. doi: 10.1016/j.arbres.2011.01.001. No abstract available. English, Spanish. PMID 21398016
- [Background] Punjabi NM, Caffo BS, Goodwin JL, Gottlieb DJ, Newman AB, O'Connor GT, Rapoport DM, Redline S, Resnick HE, Robbins JA, Shahar E, Unruh ML, Samet JM. Sleep-disordered breathing and mortality: a prospective cohort study. PLoS Med. 2009 Aug;6(8):e1000132. doi: 10.1371/journal.pmed.1000132. Epub 2009 Aug 18. PMID 19688045
- [Background] Duran Cantolla J, Esnaola Sukia S, Rubio Aramendi R, Egea Santaolalla C. [Validity of a portable recording system (MESAM IV) for the diagnosis of sleep apnea syndrome]. Arch Bronconeumol. 1994 Aug-Sep;30(7):331-8. Spanish. PMID 7952834
- [Background] Esnaola S, Duran J, Infante-Rivard C, Rubio R, Fernandez A. Diagnostic accuracy of a portable recording device (MESAM IV) in suspected obstructive sleep apnoea. Eur Respir J. 1996 Dec;9(12):2597-605. doi: 10.1183/09031936.96.09122597. PMID 8980975
- [Background] Parra O, Garcia-Esclasans N, Montserrat JM, Garcia Eroles L, Ruiz J, Lopez JA, Guerra JM, Sopena JJ. Should patients with sleep apnoea/hypopnoea syndrome be diagnosed and managed on the basis of home sleep studies? Eur Respir J. 1997 Aug;10(8):1720-4. doi: 10.1183/09031936.97.10081720. PMID 9272909
- [Background] Jimenez Gomez A, Golpe Gomez R, Carpizo Alfayate R, de la Roza Fernandez C, Fernandez Rozas S, Garcia Perez MM. [The validation of a portable 3-channel recording system (Oxyflow, Edentec) for the diagnosis of the sleep apnea syndrome]. Arch Bronconeumol. 2000 Jan;36(1):7-12. doi: 10.1016/s0300-2896(15)30226-x. Spanish. PMID 10726178
- [Background] Calleja JM, Esnaola S, Rubio R, Duran J. Comparison of a cardiorespiratory device versus polysomnography for diagnosis of sleep apnoea. Eur Respir J. 2002 Dec;20(6):1505-10. doi: 10.1183/09031936.02.00297402. PMID 12503711
- [Background] Nunez R, Rey de Castro J, Socarras E, Calleja JM, Rubio R, Aizpuru F, Duran-Cantolla J. [Validation study of a polygraphic screening device (BREAS SC20) in the diagnosis of sleep apnea-hypopnea syndrome]. Arch Bronconeumol. 2003 Dec;39(12):537-43. doi: 10.1016/s0300-2896(03)75451-9. Spanish. PMID 14636489
- [Background] Masa JF, Corral J, Pereira R, Duran-Cantolla J, Cabello M, Hernandez-Blasco L, Monasterio C, Alonso A, Chiner E, Rubio M, Garcia-Ledesma E, Cacelo L, Carpizo R, Sacristan L, Salord N, Carrera M, Sancho-Chust JN, Embid C, Vazquez-Polo FJ, Negrin MA, Montserrat JM. Effectiveness of home respiratory polygraphy for the diagnosis of sleep apnoea and hypopnoea syndrome. Thorax. 2011 Jul;66(7):567-73. doi: 10.1136/thx.2010.152272. Epub 2011 May 20. PMID 21602541
- [Background] Masa JF, Corral J, Pereira R, Duran-Cantolla J, Cabello M, Hernandez-Blasco L, Monasterio C, Alonso A, Chiner E, Zamorano J, Aizpuru F, Montserrat JM; Spanish Sleep Network. Therapeutic decision-making for sleep apnea and hypopnea syndrome using home respiratory polygraphy: a large multicentric study. Am J Respir Crit Care Med. 2011 Oct 15;184(8):964-71. doi: 10.1164/rccm.201103-0428OC. Epub 2011 Jul 7. PMID 21737584
- [Background] Kushida CA, Littner MR, Morgenthaler T, Alessi CA, Bailey D, Coleman J Jr, Friedman L, Hirshkowitz M, Kapen S, Kramer M, Lee-Chiong T, Loube DL, Owens J, Pancer JP, Wise M. Practice parameters for the indications for polysomnography and related procedures: an update for 2005. Sleep. 2005 Apr;28(4):499-521. doi: 10.1093/sleep/28.4.499. PMID 16171294
- [Background] Duran Cantolla J, Amilibia Alonso J, Barbe Illa F, Capote Gil F, Gonzalez-Mangado N, Jimenez Gomez A, Marin Trigo JM, Masa Jimenez JF, Montserrat Canal JM, Teran Santos J. [Availability of technical resources for diagnosis and treatment of sleep obstructive apnea syndrome in state hospitals in Spain]. Arch Bronconeumol. 1995 Nov;31(9):463-9. No abstract available. Spanish. PMID 8520819
- [Background] Johns MW. Daytime sleepiness, snoring, and obstructive sleep apnea. The Epworth Sleepiness Scale. Chest. 1993 Jan;103(1):30-6. doi: 10.1378/chest.103.1.30. PMID 8417909
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Netzer NC, Stoohs RA, Netzer CM, Clark K, Strohl KP. Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome. Ann Intern Med. 1999 Oct 5;131(7):485-91. doi: 10.7326/0003-4819-131-7-199910050-00002. PMID 10507956
- [Background] Ragette R, Wang Y, Weinreich G, Teschler H. Diagnostic performance of single airflow channel recording (ApneaLink) in home diagnosis of sleep apnea. Sleep Breath. 2010 Jun;14(2):109-14. doi: 10.1007/s11325-009-0290-2. Epub 2009 Aug 28. PMID 19714380